CLINICAL TRIAL: NCT01902680
Title: Phase II Study of Feasibility of Focal Therapy for Prostate Cancer of Good Prognosis With Permanent I125 Localized Implant.
Acronym: CURIEFOCALE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12 URO 06
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Localized Prostate Cancer
Keywords: Prostate cancer, permanent implant brachytherapy, image fusion, focal therapy, active surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal brachytherapy (Experimental): Focal brachytherapy with permanent I125 localized implant.
  Interventions: Radiation: Focal brachytherapy

INTERVENTIONS:
Radiation: Focal brachytherapy — Focal brachytherapy with permanent I125 localized implant.

SUMMARY:
This is a pilot prospective biomedical study of interventional type which includes 17 patients on 24 months (12 months of inclusion and 12 months of follow-up).

The objective of this study is to verify that the focal therapy technique used (with the help of Koelis® system) allows to obtain optimal dosimetric coverage of the prostate target (ie dose of 160 Gy +-5% delivered on the envelope isodose) evaluated by CT scan performed 30 days after implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Men of more than 18 years old
2. Patient with localized prostate cancer with a good prognosis (AMICO classification), ie satisfying the following conditions according to the urologist medical record transmitted:

   * Lesion classified T1c or T2a based on digital rectal exam
   * histologically proven diagnosis of prostatic adenocarcinoma with a Gleason score ≤ 6
   * Serum Prostatic Specific Antigen (PSA) <10ng/ml
3. Patient for whom the Multidisciplinary Consultative Meeting (RCP) has adopted the following treatment options: active surveillance, brachytherapy, radical prostatectomy or external radiation
4. Patient with good micturating function at inclusion, defined by IPSS score <10 (IPSS Questionnaire)
5. Patient for whom the result of centralized PSA assay confirms a serum level < 10ng/ml
6. Patient for whom the unique and intracapsular character of the target area (area to be treated) was confirmed on pre implantation multimodal MRI imaging (ESUR Score ≥ 9) and whose major axis has a size ≤ 20 mm
7. Patient with a Gleason score on the target ≤ 6 (3 +3) confirmed on biopsies performed using KOELIS ® system and with no other derogatory criteria such as the invasion of the entire core or the presence of a grade 4 or perineural emboli
8. Patients without history of transurethral resection that could have significantly modified the anatomy of the gland nor obstructive adenoma
9. Patient who accepts, at the end of the study, the principle of active surveillance for the rest of the gland and the treated area according to the current standard protocol
10. WHO ≤ 2
11. Patient with life expectancy > 10 years
12. Informed consent obtained and signed before any specific procedure in the study
13. Patient affiliated to social security regimen

Exclusion Criteria:

1. Image in favour of the crossing of the capsule, based on pre-implantation multimodal MRI (stage T2 MRI only)
2. Image in favor of the invasion of the seminal vesicle, based on pre-implantation multimodal MRI (stage T2 MRI only)
3. Multifocal lesions (ESUR ≥ 9/15) to the pre-implantation multimodal MRI and for which biopsies have shown the cancerous nature
4. Lesion with larger diameter ≥ 20mm, to the pre-implantation multimodal MRI
5. Patient who requires pre-implantation hormonal treatment in order to reduce prostatic volume
6. Patient with current indication against prostate brachytherapy, including a significant limitation of the mobility of the hips, a prostate volume greater than 60 cm3 (measured by planimetry MRI) or a significant dysuria (IPSS ≥ 10)
7. Patient unable to follow procedures, visits, examinations described in the the study
8. Patient with absolute indication against imaging tests (significant claustrophobia, wearing a heart valve, pacemaker, ..)
9. Man of childbearing age who do not want follow the instructions about sexual activities and condom use during the days following the treatment of brachytherapy and / or unwilling to hold (him or her partner) effective contraception for the duration of the study
10. Any concomitant or previous malignant disease in the past five years with the exception of superficial basal cell carcinoma or non-metastatic of the skin
11. Any prior systemic chemotherapy within 5 years prior to inclusion for malignant disease in the medical history
12. Any coexisting medical condition that in the opinion of the investigator could be a risk in this study
13. Patient protected by law

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08-23 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of focal therapy will be evaluated with dosimetric study by CT scan / MRI performed 30 days after implantation | 3 years
  Feasibility of focal therapy will be evaluated in terms of "success" or "failure" : success will be obtained in case of delivered dose of at least 152 Gy on the 1st dose enveloping the Planning Target Volume, evaluated on CT scan/MRI performed at Day 30

SECONDARY OUTCOMES:
Progression-free-survival according to Phoenix criterion | 3 years
  Progression-free-survival is defined as the time from patient inclusion to the date of biological progression according to Phoenix criterion
Quality of life study using 3 Patient questionnaires | 3 years
  Quality of life will be evaluated using 3 Patient questionnaires : the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ)C30 Questionnaire, the International Index of Erectile Function Questionnaire and the International Prostate Symptom Score Questionnaire
Absence of tumor residuals in the target treated zone | 3 years
  The absence of tumor residuals in the target treated zone will be evaluated on on biopsies performed 1 year after implantation
Toxicity evaluation | 3 years
  Toxicity will be evaluated according to the classification of NCI Common Toxicity Criteria for Adverse Effects (CTCAE) V4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius REGAUD, Toulouse, France